CLINICAL TRIAL: NCT01571089
Title: Anxiety Treatment Inspired by Dialectical Behavior Therapy (DBT) - An Alternative for Patients Who Previously Received Exposure-based Treatment for Anxiety Without Sustained Improvements.
Brief Title: Anxiety Treatment Inspired by Dialectical Behavior Therapy (DBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Sara Edlund, Doctoral student & Clinical psychologist, Örebro County Council
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLL-189011
Record Dates: First submitted 2012-03-26; First posted 2012-04-04 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Treatment Resistant Anxiety Disorders
Keywords: Dialectical behavior therapy; cognitive behavioral therapy; emotion regulation; emotion dysregulation; anxiety disorders; skills training
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBT-inspired exposure treatment (Experimental): DBT-inspired exposure treatment.
  Interventions: Behavioral: DBT-inspired anxiety treatment

INTERVENTIONS:
Behavioral: DBT-inspired anxiety treatment — In short, the treatment is 24 sessions consisting of skills-training strategies and exposure strategies. The idea is that the patient during the treatment will learn and practice the skills needed to handle exposures.

SUMMARY:
The main interest in this study is to investigate if it is possible to use strategies from Dialectical Behavior Therapy (DBT) to increase effectiveness of ordinary Cognitive Behavioral Therapy (CBT) for patients with anxiety disorders. For the patients included in this study, previous exposure-based treatment should have been unsuccessful (drop-out, relapse or lack of positive results after treatment).

ELIGIBILITY:
Inclusion Criteria:

* Currently diagnosed with an anxiety disorder. To be included, the level of anxiety in a critical situation should be high and of a more acute type, unlike the lower more generalized anxiety in for example generalized anxiety disorder.
* Previous exposure-based treatment should have been unsuccessful (drop-out, relapse or lack of positive results after treatment).

Exclusion Criteria:

* Severe depression.
* Psychotic disorder.
* A documented neuropsychiatric diagnosis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in anxiety (Clark, D. M., Ehlers, A., McManus, F., Hackmann, A., Fennell, M., Campbell, H., Flower, T., Davenport, C., Louis, B., 2003). | Every day during baseline phase, an expected average of 3 weeks. Everyday during treatment, an expected duration of 24 weeks. Everyday during 6 mo. follow-up, an expected average of 3 weeks.
  A modified 6-item questionnaire measuring changes in different aspects of anxiety during the day. Originally developed to measure social anxiety.

SECONDARY OUTCOMES:
Positive Negative Affect Scale (PANAS), (Watson, Clark & Tellegan, 1988). | Once a week during baseline phase, an expected average of 3 weeks. Once a week during treatment, an expected duration of 24 weeks. Once a week during 6 mo. follow-up, an expected average of 3 weeks.
  A 20-item questionnaire measuring positive and negative affect during the past week. The questionnaire is used to evaluate changes in positive and negative affect.
Overall Anxiety Severity and Impairment Scale (OASIS), (Barlow, 2011). | Once a week during baseline phase, an expected average of 3 weeks. Once a week during treatment, an expected duration of 24 weeks. Once a week during 6 mo. follow-up, an expected average of 3 weeks.
  A 5-item questionnaire measuring different aspects of anxiety during the past week. The questionnaire is used to evaluate changes in anxiety symtoms.
Overall Depression Severity and Impairment Scale (ODSIS), (Barlow, 2011). | Once a week during baseline phase, an expected average of 3 weeks. Once a week during treatment, an expected duration of 24 weeks. Once a week during 6 mo. follow-up, an expected average of 3 weeks.
  A 5-item questionnaire measuring different aspects of depression during the past week. The questionnaire is used to evaluate changes in depressive symtoms.
Difficulties in Emotion Regulation Scale (DERS), (Gratz & Roemer, 2004). | Five times total. Pre baseline, post baseline/post treatment, after 14 weeks of treatment, post treatment and at 6 mo. follow-up.
  A 36-item self-report instrument that measure changes in difficulties in emotion regulation.
Five Fazet Mindfulness Questionnaire (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). | Five times total. Pre baseline, post baseline/post treatment, after 14 weeks of treatment, post treatment and at 6 mo. follow-up.
  A 39-item questionnaire measuring changes in different aspects of mindfulness.
WHOQOL-BREF (Skevington, Lofty, O´Connel & WHOQOL Group, 2004). | Five times total. Pre baseline, post baseline/post treatment, after 14 weeks of treatment, post treatment and at 6 mo. follow-up.
  A 26-item self-report instrument that measure changes in quality of life.
Structured Clinical Interview for DSM-IV-I (SCID-I), (First, Spitzer, Gibbon, & Williams, 2001). | Pre- and post treatment
  A structural interview assessing axis-I disorders. This instrument is used to evaluate changes in axis-I disorders in the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Clinic, Hallsberg, Örebro County, Sweden